CLINICAL TRIAL: NCT00946309
Title: In Vivo Effects of Sulforaphane Supplementation on Normal Human Prostate
Brief Title: Effects of Sulforaphane on Normal Prostate Tissue
Acronym: PHASE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Seattle Institute for Biomedical and Clinical Research (Other); Johns Hopkins University (Other); University of Washington (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Lin, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PHS 2333.00; 6969 (Other: FHCRC)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Sulforaphane Extract (Experimental)
  Interventions: Drug: High Sulforaphane Extract (Broccoli Sprout Extract)
- Placebo (Placebo Comparator)
  Interventions: Drug: Microcrystalline Cellulose NF (placebo)

INTERVENTIONS:
Drug: High Sulforaphane Extract (Broccoli Sprout Extract) — 100 umol sulforaphane, every other day for 5 weeks
  Other Names: Broccoli Sprout Extract
  Arms: High Sulforaphane Extract
Drug: Microcrystalline Cellulose NF (placebo) — 250 mg every other day for 6 weeks
  Arms: Placebo

SUMMARY:
The investigators proposed to identify the biological effects of a high-sulforaphane broccoli sprout extract in normal prostate tissue.

The investigators hypothesize that consumption of high-sulforaphane broccoli sprout extract every other day will inhibit growth of prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40-75 years
* Low or intermediate grade prostate cancer (as defined by Gleason sum less than or equal to 7) and clinical stage T1 or T2
* Serum Prostate specific antigen less than 20 ng/ml
* Have elected radical prostatectomy, Brachytherapy or active surveillance as their primary treatment

Exclusion Criteria:

* No current physician diagnosed disease (including but not limited to): kidney disease requiring dialysis, cognitive deficits, substance abuse
* BMI < 18.5 kg/m2 or > 40 kg/m2
* Use of any hormonal treatments, including but not limited to testosterone
* Any previous cancer diagnosis or treatment within the previous five years, excluding non-melanoma skin cancer
* Inability or unwillingness to eat a diet that is free of Brassica vegetables for the duration of the study
* Use of any dietary supplements other than a multivitamin (including herbal preparations)
* Allergy to cruciferous vegetables or any of the specific fillers used in the placebo
* Usual consumption of > 5 servings per week of Brassica vegetables

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Lin, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- VA Puget Sound, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from July 2010 to April 2014 at the VA Puget Sound Health Care System.
Pre-assignment Details: There were no pre-assignment events. Group assignment occurred at the time of participant enrollment.
Groups:
- Sulforaphane: High Sulforaphane Extract (Broccoli Sprout Extract): 100 umol sulforaphane, every other day for 5 weeks
- Placebo: Microcrystalline Cellulose NF (placebo): 250 mg every other day for 5 weeks
Period: Overall Study
Arm/Group | Sulforaphane | Placebo
Started | 22 | 23
Completed | 21 | 19
Not Completed | 1 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Procedure cancelled/discontinued | 0 | 3

BASELINE CHARACTERISTICS:
Population: One participant enrolled to the placebo arm was determined to be ineligible, and was withdrawn from the study Two additional participants enrolled to the placebo arm became ineligible after enrollment, and were withdrawn from the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulforaphane | Placebo | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 29
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (5.4) | 62.8 (4.3) | 62.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 16 | 20 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Gene Expression of Phase II Enzymes
Description: Change in Phase II enzyme expression
Time Frame: Baseline and 5 weeks
Population: Due to budget restrictions, outcome data from only collected from the first 20 participants
Measure: Mean (Standard Deviation); unit: -fold change in expression
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 10 | 10
-fold change in expression
  Glutathione peroxidase 4 (GPX4) expression | -0.36 (2.0) | 0.26 (1.1)
  Glutathione S-transferase A2 (GSTa2) expression | 0.15 (4.1) | -0.59 (3.0)
  NAD(P)H:quinone oxidoreductase (NQ01) expression | -0.02 (1.3) | 0.42 (0.10)
  RODH5 F2/R2 expression | -0.10 (2.6) | -0.02 (2.6)
  Superoxide dismutase (SOD1) expression | 0.35 (1.1) | 0.5 (1.0)

2. Primary Outcome: Lipid Oxidation
Description: Blood F2 Isoprostane levels
Time Frame: Baseline and 5 weeks
Population: Outcome data were not collected due to budget restrictions
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: DNA Oxidation
Description: Prostate tissue 8-hydroxy-2'-deoxyguanosine (8OHdG) levels
Time Frame: Five weeks
Population: Outcome data were not collected due to budget restrictions
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: DHT Levels
Description: Change in serum dihydrotestosterone (DHT) levels
Time Frame: Baseline and 5 weeks
Population: Due to budget restrictions, outcome data from only collected from the first 25 participants
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 13
pg/mL | 2.09 (77.8) | 19.33 (98.0)

5. Primary Outcome: Testosterone Levels
Description: Change in testosterone (T) levels
Time Frame: Baseline and 5 weeks
Population: Due to budget restrictions, outcome data from only collected from the first 25 participants
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 13
ng/dL | -36.79 (79.1) | 5.75 (156.8)

6. Primary Outcome: 3-alpha-diol Gluconate Levels
Description: Change in serum 3-alpha-diol gluconate(3α-DG) levels
Time Frame: Baseline and 5 weeks
Population: Due to budget restrictions, outcome data from only collected from the first 25 participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sulforaphane | Placebo
Number analyzed (Participants) | 12 | 13
ng/mL | -0.69 (1.6) | 0.39 (1.2)

ADVERSE EVENTS:
Description: Participants were asked to report the frequency/severity of gastrointestinal-related symptoms weekly.
  Adverse event data for the sulforaphane arm is based only on 21 because all data/specimens for one participant (who was ineligible and mistakenly enrolled) was destroyed per Institutional Review Board regulations.
Arm/Group | Sulforaphane | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 19/21 | 18/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulforaphane (N=21) | Placebo (N=23)
Burping (Grade 1) (Gastrointestinal disorders) | 4 (8) | 6 (6) — Grade 1: Symptomatic but not interfering with activities of daily living daily living
Burping (Grade 2) (Gastrointestinal disorders) | 1 (3) | 0 (0) — Grade 2: Symptomatic and interfering with activities of
Abdominal Bloating (Grade 1) (Gastrointestinal disorders) | 5 (6) | 3 (3) — Grade 1: No change in bowel function or oral intake
Abdominal bloating (Grade 2) (Gastrointestinal disorders) | 1 (3) | 0 (0) — Grade 2: Symptomatic decreased oral intake; change in bowel function
Heartburn (Grade 1) (Gastrointestinal disorders) | 5 (9) | 3 (3)
Heartburn (grade 2) (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (7) | 4 (4)
Vomiting (Grade 1) (Gastrointestinal disorders) | 1 (3) | 3 (3)
Vomiting (Grade 2) (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal Pain (Grade 1) (Gastrointestinal disorders) | 5 (5) | 2 (4)
Abdominal Pain (Grade 2) (Gastrointestinal disorders) | 1 (2) | 2 (4)
Flatulence (Grade 1) (Gastrointestinal disorders) | 9 (17) | 4 (7)
Flatulence (Grade 2) (Gastrointestinal disorders) | 2 (5) | 2 (3)
Diarrhea (Grade 1) (Gastrointestinal disorders) | 6 (8) | 7 (11)
Constipation (Grade 1) (Gastrointestinal disorders) | 3 (3) | 4 (11)
Constipation (Grade 2) (Gastrointestinal disorders) | 3 (7) | 0 (0)
Change in Stool Consistency (Grade 1) (Gastrointestinal disorders) | 0 (0) | 4 (11)
Increase in Appetite (Gastrointestinal disorders) | 0 (0) | 2 (4)
Hyperglycemia (Grade 3) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Light Headed (Grade 1) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Grade 1) (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No